CLINICAL TRIAL: NCT06254326
Title: ADAGiO: Adoptive Cellular Therapy for the TreAtment of Recurrent OliGodendrogliOma (OG) Adult Patients
Acronym: ADAGiO
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Oligo Nation, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB202301855; OCR44817 (Other: University of Florida)
Record Dates: First submitted 2024-01-22; First posted 2024-02-12 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Oligodendroglioma; Progressive Oligodendroglioma
Keywords: Immunotherapy; Brain Tumor
MeSH Terms: conditions — Oligodendroglioma; Brain Neoplasms | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; Diphtheria-Tetanus Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Adoptive Cellular Therapy (Experimental): All participants will receive 9 intradermal DC vaccines (three -bi-weekly (q2 weeks) for priming, monthly for additional 2-3 cycles during T cell expansion, and three bi-weekly during T cell engraftment), a single i.v. infusion of ex vivo expanded tumor-reactive T cells, and a i.v. single infusion of autologous HSCs.
  Interventions: Biological: TTRNA-DC vaccines with GM-CSF; Biological: Autologous Hematopoietic Stem cells (HSCs); Biological: TTRNA-xALT; Drug: Td vaccine

INTERVENTIONS:
Biological: TTRNA-DC vaccines with GM-CSF — Participants will receive up to 9 intradermal DC vaccines (three -bi-weekly (q2 weeks) for priming, monthly for additional 2-3 cycles during T cell expansion, and three bi-weekly during T cell engraftment
Biological: Autologous Hematopoietic Stem cells (HSCs) — Participants will receive a single infusion of autologous CD34+ HSCs
Biological: TTRNA-xALT — Participants will receive a single infusion of ex vivo expanded tumor-reactive T cells
Drug: Td vaccine — All patients will receive a full Td booster IM vaccine 4-24 hours prior to Vaccine #1 and vaccine site pretreatment with a one-fifth dose of Td intradermally, at the site of planned vaccine, 4-24 hours prior to vaccines #3, #5, #7 and #9.

SUMMARY:
This study will enroll 6 DLT evaluable subjects (up to 12 patients total) where we will evaluate feasibility and safety of adoptive cellular therapy combined with IDH1/2 inhibitors in patients with recurrent or progressive oligodendroglioma WHO grade 2 and WHO grade 3.

DETAILED DESCRIPTION:
After screening consent, subjects will undergo standard of care resection or biopsy for confirmatory diagnosis of disease progression and aseptic collection of tumor material for DNA and RNA extraction and sequencing, amplification, and loading of autologous DCs. Following biopsy and confirmatory pathologic diagnosis, eligible patients will be enrolled in treatment.

After surgery, patients will undergo a G-CSF mobilized pheresis to collect PBMCs for DC generation and CD34+ HSCs. Amplified tumor RNA obtained from surgically resected or biopsied specimens will be used to generate total tumor RNA-pulsed DCs (TTRNA-DCs) manufactured while patients initiate salvage chemotherapy regimen after surgery.

Salvage chemotherapy with IDH1/2 inhibitor will initiate 1-2 weeks after G-CSF mobilized leukapheresis for 1-3 cycles after which, treatment cycles will be paused, and the patients will receive 3 priming TTRNA-DCs vaccines every 2 weeks and undergo a non-mobilized leukapheresis to collect vaccine-boosted lymphocytes for ex vivo T cell expansion and generation of additional TTRNA-DC vaccines. Treatment with IDH1/2 inhibitor will resume with monthly TTRNA-DC vaccines for an additional 1-3 cycles until ex vivo expanded T cells are manufactured.

For ACT, patients will undergo non-myeloablative conditioning with cyclophosphamide /fludarabine. The total immunotherapy regimen will consist of up to 9 intradermal DC vaccines (three -bi-weekly (q2 weeks) for priming, monthly for additional 2-3 cycles during T cell expansion, and three bi-weekly during T cell engraftment), a single i.v. infusion of ex vivo expanded tumor-reactive T cells, and a i.v. single infusion of autologous HSCs.

The duration of treatment from enrollment to completion of DLT window is anticipated to be 7 to 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 years and above
* Tumor tissue obtained on a screening consent is available.
* Confirmed with recurrent/progressive IDH-mutant 1p/19q co-deleted Oligodendroglioma WHO grade 2 or WHO grade 3, more than 12 weeks from completion of radiation.
* Karnofsky Performance Status ≥ 60
* Must be a candidate for surgery/biopsy
* Adequate bone marrow and organ function as defined below:

  * ANC ≥ 1,000/mcL
  * Platelets ≥ 100,000/mcL
  * Hemoglobin ≥ 9 g/dL (can be transfused)
  * Serum creatinine ≤ 1.5 x IULN OR Creatinine clearance by Cockcroft-Gault ≥ 60 mL/min for patients with serum creatinine > 1.5 x IULN
  * Serum total bilirubin ≤ 1.5 x IULN OR Direct bilirubin ≤ IULN for patients with total bilirubin > 1.5 x IULN
  * AST (SGOT) and ALT (SGPT) ≤ 3 x IULN
* For females of childbearing potential, negative serum pregnancy test at enrollment
* For women and men of childbearing potential (WOCBP) must be willing to use acceptable contraceptive methods

Exclusion Criteria:

* Disease progression during treatment with an anti-IDH-1 or anti IDH-2
* Prior invasive malignancy (except for non-melanomatous skin cancer) unless disease free for ≥ 3 years.
* Metastases detected below the tentorium or beyond the cranial vault and leptomeningeal involvement.
* Multifocal disease.
* Corticosteroids equivalent to ≥ 4mg dexamethasone daily.
* HIV, Hepatitis B, or Hepatitis C seropositive.
* Known active infection or immunosuppressive disease.
* Autoimmune disease requiring medical management with immunosuppressant.
* Pregnancy or lactation, due to possible adverse effects on the developing fetus or infant.
* Treatment with another investigational drug or other intervention within 30 days prior to projected first dose of study treatment (Priming phase with TTRNA-DC).
* Severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization.
  * Transmural myocardial infarction within the last 6 months.
  * Acute bacterial or fungal infection requiring intravenous antibiotics at time of enrollment.
  * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy.
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects.
  * Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive.
  * Major medical illnesses or psychiatric impairments that, in the investigator's opinion, will prevent administration or completion of protocol therapy.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Prevalence of enrolled subject who receive qualified immunotherapy investigational product. | enrollment up to 9 months
  Feasibility will be measured by the number of patients who receive autologous dendritic cells, T cells and hematopoietic stem cells that meet the FDA IND defined quality assurance and quality control release criteria. A minimum of 66.7% of enrolled subject must achieve this criterion for feasibility endpoint.
Incidence of investigational treatment related severe toxicity (Dose-limiting toxicity event) assessed during the period beginning with administration of ex vivo expanded TTRNA T cells through 6 weeks post infusion. | enrollment to completion of DLT window; up to 9 months.
  Safety will be defined as < 1 DLT out of six enrolled and treated subjects during the defined period of administration of ex vivo expanded TTRNA T cells through 6 weeks post infusion. Investigational treatment related CTCAE V5.0 adverse events 1) Grade III or greater non-neurologic toxicity; 2) Grade III neurologic toxicity that does not improve to Grade II or better within 5 days; or 3) Grade IV neurologic toxicity will be recorded toward DLT.

CONTACTS AND LOCATIONS:
Overall Officials: Duane Mitchell, MD, PhD, Study Chair — University of Florida; Ashley Ghiaseddin, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Health Shands Hospital, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No